CLINICAL TRIAL: NCT07023172
Title: Multicenter, Prospective, Observational Study on the Treatment of Type 2 Diabetes With Proline Plus Empagliflozin Tablets
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HDHYJ-LC-1
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Proline plus empagliflozin tablets
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a post-marketing, multicenter, prospective, observational study designed to evaluate the efficacy and safety of Proline Plus Empagliflozin Tablets in the real-world clinical treatment of type 2 diabetes mellitus. The study does not interfere with routine clinical practice, and Proline Plus Empagliflozin Tablets may be used either as monotherapy or in combination with other therapeutic agents based on actual clinical needs.

DETAILED DESCRIPTION:
This study is a post-marketing study aimed at evaluating the effectiveness and safety of proline-containing gliflozin tablets in the real-world clinical treatment of type 2 diabetes mellitus. The study is designed as a multicenter, prospective, observational study. This research does not interfere with clinical diagnosis and treatment, and proline-containing gliflozin tablets may be used as monotherapy or in combination with other therapeutic drugs based on actual needs.

Dosage and administration of proline-containing gliflozin tablets:

For newly diagnosed type 2 diabetes patients: The initial dose is one tablet once daily, taken with meals. For patients requiring enhanced glycemic control who tolerate 25 mg once daily, the dose may be increased to 50 mg once daily, taken with meals.

This study includes a screening period (D-14 to D0) and a treatment period (12 weeks ± 7 days, 24 weeks ± 28 days, 48 weeks ± 28 days), totaling 4 visit points. During the study, patients may undergo examinations based on actual clinical needs. The trial requires recording patients' baseline physical examinations, study drug prescription and concomitant medication use, examinations performed according to clinical needs, and the occurrence of adverse events or adverse drug reactions.

The EQ-5D score will be assessed for all subjects. Additionally, for subjects aged 50 years or older (with an education level of elementary school or above), the MoCA (Version 7.1) score and cognitive impairment assessment will be conducted at all visit points except the second one.

Subgroups will be defined based on baseline age (<65 years, ≥65 years), HbA1c (HbA1c ≥7%, ≥9%, or ≥11%), BMI (BMI <24.0 kg/m², 24.0 kg/m² ≤ BMI ≤ 28.0 kg/m², BMI ≥28.0 kg/m²), and concomitant medications (number and types of glucose-lowering drugs) to observe differences in efficacy between subgroups.Subgroups will also be defined based on comorbidities to observe the glucose-lowering efficacy and changes in relevant clinical indicators in different comorbidity populations, such as:Chronic kidney disease population: Focus on changes in serum creatinine (SCr), urine protein (Pro), estimated glomerular filtration rate (eGFR), urine albumin-to-creatinine ratio (UACR), and major adverse kidney events (MAKE).Cardiovascular disease population: Focus on major adverse cardiovascular events (MACE) and echocardiographic indicators.

Retinopathy population: Focus on fundus examination results.Cognitive impairment population: Focus on changes in MoCA scores.The analysis indicators will be based on actual analyzable data generated during the study.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥18 years, regardless of gender. 2.Clinically diagnosed with type 2 diabetes mellitus (per the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes Mellitus [2020 Edition]).

  3.Deemed suitable by the investigator for treatment with proline-containing gliflozin tablets (Hui You Jing) and being prescribed this medication for the first time.

  4.Availability of glycated hemoglobin (HbA1c) test results within 4 weeks prior to enrollment.

  5.Voluntary participation with signed informed consent.

Exclusion Criteria:

- 1.History of moderate to severe renal impairment (eGFR <30 mL/min/1.73 m²), end-stage renal disease, or dialysis.

2.Acute or chronic metabolic acidosis, including diabetic ketoacidosis. Severe allergy to gliflozin or any excipient of the study drug. 3.Current or recent (within 1 month) participation in any other clinical trial. 4.Investigator judgment of unsuitability for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥18 years, no gender restriction; clinically diagnosed with type 2 diabetes mellitus (per Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes Mellitus [2020]); deemed by investigators as suitable for and initiating empagliflozin treatment for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
HbA1c <7.0% | at 24 weeks
  Glycemic control rate at 24 weeks, where glycemic control is defined as HbA1c <7.0%

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xinyang Central Hospital, Xinyang, Henan
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu